CLINICAL TRIAL: NCT00001047
Title: An Open-Label, Randomized Trial of Four Treatment Regimens for Patients With Disseminated Mycobacterium Avium Complex Disease and Acquired Immunodeficiency Syndrome (AIDS)
Brief Title: Study of Four Different Treatment Approaches for Patients Who Have Mycobacterium Avium Complex Disease (MAC) Plus AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CPCRA 027; 11577 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Clofazimine; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Clarithromycin; Clofazimine; Rifabutin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Clofazimine
Drug: Rifabutin

SUMMARY:
To compare the safety and efficacy of two doses of clarithromycin in combination with ethambutol and either rifabutin or clofazimine for the treatment of disseminated Mycobacterium avium Complex (MAC) disease in AIDS patients.

Recommendations have been issued for AIDS patients with disseminated MAC to be treated with at least two antimycobacterial agents and for every regimen to include a macrolide (clarithromycin or azithromycin). However, the optimal treatment for disseminated MAC remains unknown.

DETAILED DESCRIPTION:
Recommendations have been issued for AIDS patients with disseminated MAC to be treated with at least two antimycobacterial agents and for every regimen to include a macrolide (clarithromycin or azithromycin). However, the optimal treatment for disseminated MAC remains unknown.

Patients are randomized to receive clarithromycin at one of two doses plus ethambutol and either rifabutin or clofazimine. Patients are followed at 1, 2, and 4 months and every 4 months thereafter for a minimum of 1.5 years to a common closing date.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended in patients with CD4 count <= 200 cells/mm3:

* Antiretroviral therapy.
* PCP prophylaxis.

Allowed in all patients:

* Isoniazid preventive therapy.

Patients must have:

* HIV infection.
* Evidence of disseminated MAC infection.

NOTE:

* Pregnant women are permitted to enroll following counseling by their clinician regarding the potential negative side effects of the study medications. These drugs should be used in pregnancy only when the potential benefits outweigh the risks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to the study drugs.
* Other concurrent mycobacterial disease requiring therapy, i.e., disseminated nontuberculous mycobacterial infection or active tuberculosis.

Concurrent Medication:

Excluded:

* Additional medications with antimycobacterial activity (unless patient is failing or intolerant of assigned study regimen).
* Drugs with potential additive toxicity or with potential interaction with study drugs (e.g., fluconazole).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Study Completion 1996-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cohn D, Study Chair; Fisher E, Study Chair; Horsburgh CR, Study Chair
Locations (16):
- United States (16):
  - Community Consortium of San Francisco, San Francisco, California
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Baltimore Trials, Baltimore, Maryland
  - Comprehensive AIDS Alliance of Detroit, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners Research, Albuquerque, New Mexico
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - Portland Veterans Adm Med Ctr / Rsch & Education Grp, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Cohn DL, Fisher EJ, Peng GT, Hodges JS, Chesnut J, Child CC, Franchino B, Gibert CL, El-Sadr W, Hafner R, Korvick J, Ropka M, Heifets L, Clotfelter J, Munroe D, Horsburgh CR Jr. A prospective randomized trial of four three-drug regimens in the treatment of disseminated Mycobacterium avium complex disease in AIDS patients: excess mortality associated with high-dose clarithromycin. Terry Beirn Community Programs for Clinical Research on AIDS. Clin Infect Dis. 1999 Jul;29(1):125-33. doi: 10.1086/520141. PMID 10433575